CLINICAL TRIAL: NCT04336033
Title: Validation and Evaluation of a Newly Developed Mobile Diet App for Enhancing Dietary Adherence for Patients With Chronic Kidney Disease (CKD)
Brief Title: Validation and Evaluation of a Newly Developed Mobile Diet App
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Jazlina binti Syahrul, Principle Investigator [Dietitian], Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NMRR-19-3569-50972
Record Dates: First submitted 2020-03-19; First posted 2020-04-07 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Diseases; Chronic Kidney Disease stage3; Chronic Kidney Disease stage4; Chronic Kidney Disease Stage 5; Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: MyNutriKidney
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: A 12-week, open-label, multicenter, randomized controlled pilot study (RCT) will be implemented to evaluate the feasibility, acceptability as well as preliminary efficacy of the newly developed renal diet app in enhancing dietary adherence among CKD patients at different stages in Malaysia. Participants will be randomly assigned in the ratio of 1:1 into two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counseling + Renal Diet App (Experimental): Subjects in the intervention group will receive an individualized dietetic counseling from the researcher aided with the newly developed renal diet app for educative purpose and aiding tool to enhance the dietary adherence among CKD patients
  Interventions: Other: Counseling; Other: Renal Diet App
- Counseling + Printed Nutrition Pamphlet (Placebo Comparator): Individualized dietetic counseling aided with printed nutrition pamphlet prepared by Ministry of Health, Malaysia
  Interventions: Other: Counseling; Other: Printed Nutrition Pamphlet

INTERVENTIONS:
Other: Counseling — Subjects in the both arms will receive individualized dietetic counseling as the standard dietetic care in Malaysia
Other: Renal Diet App — Individualized dietetic counseling aided with a newly developed renal diet app for educative purpose and aiding tool to enhance the dietary adherence among CKD patients. Training on the use of the app will be provided to the subjects prior to the commencement of the intervention. Subjects will be trained on the use of the home screen, icons, feedback screens, the process of entering dietary and fluid intake data and selecting portion sizes. Subjects are considered as competent users when they could correctly record the foods and drinks with correct portion size eaten in the past 24 hours and successfully save the data.
  Other Names: MyNutriKidney
  Arms: Counseling + Renal Diet App
Other: Printed Nutrition Pamphlet — After the counseling session, a standardized renal nutrition pamphlet prepared by dietitians from Universiti Putra Malaysia and Hospital Serdang will be given for patient's educative purpose.
  Since the mobile application is intended for patient's education and self-monitoring (food diary) purposes, and thus, to ensure the comparability between intervention and control groups, the patients in control group will be trained to record their diet intakes manually using the recommended approach 3-day diet records. Nutritional feedback or advices on the diet records will be given to the participants during follow up sessions.
  Arms: Counseling + Printed Nutrition Pamphlet

SUMMARY:
A 12-week, prospective, multicenter, open-label pilot randomized controlled trial (RCT) will be carried out to determine the feasibility, acceptability and potential clinical efficacy of a newly developed mobile diet app among CKD populations at different stages in Malaysia. Participants will be randomly assigned into either (i) intervention group (mobile diet app) or (ii) control group (dietary counseling using conventional pamphlet).

DETAILED DESCRIPTION:
General Objective: To evaluate a newly developed mobile diet app in enhancing dietary adherence for patients with chronic kidney disease.

Specific Objectives:

1. To validate the newly developed mobile diet app for patient with chronic kidney disease.
2. To determine the feasibility and acceptability of this newly developed mobile diet app among patients with chronic kidney disease.
3. To evaluate the preliminary efficacy of the newly developed mobile diet app in enhancing dietary adherence in patients with chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed CKD / eGFR < 60 ml/min/1.73m2 for ≥ 3 months (only applicable to pre-dialysis patients.
2. Undergone maintenance dialysis for at least 3 months (only applicable to dialysis patients)
3. Possessing smartphone and is willing to use health app
4. Alert and oriented
5. At least 18 years of age

Exclusion Criteria:

1. Inability to use the smartphone app (e.g. due to vision problems)
2. Hard to comply with home monitoring (e.g. suffering from anxiety or depression)
3. Refuse to comply with dietary prescription
4. Patients who participate in other study at the same time
5. Patients who have participated in another research study involving an investigational product in the past 12 weeks preceding enrollment.
6. Planning for kidney transplant over the study duration.
7. Female patients who are pregnant, lactating or planning a pregnancy during the course of the trial.
8. Participants who are receiving nutritional support (i.e. enteral and intra-venous route).
9. Participants who are currently receiving active treatment for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (eGFR) | 3 months
  Estimated glomerular filtration rate (eGFR) will be recorded in of mL/min/1.73m2.
Serum Kidney Function Test | 3 months
  Routine collected biochemical results from the patients' medical records:
  - urea, sodium, chloride, potassium and creatinine will be measured in mmol/L
Serum Hemoglobin A1C Test | 3 months
  Routine collected biochemical results from the patients' medical records for HbA1C (%)
Serum Blood Sugar Profile | 2 weeks
  Routine collected biochemical results from the patients' medical records and blood sugar (mmol/L) also will be recorded if patient had done self-monitoring blood glucose at home
Albuminuria | 12 weeks
  Routine collected urine analysis to measure urine albumin (mg) if there is presence of albumin or protein
Dietary History | 6 weeks
  Three-day diet records (3DDR) : 2 days weekdays + 1 weekend / dialysis and non-dialysis day. Measured unit is in kilocalories (kcal)/day
Dietary Adherence | 6 weeks
  End Stage Renal Disease Adherence Questionnaire (ESRD-AQ):
  - validated questionnaires which consists of 4 subscales pertaining dialysis, medication, dietary and fluid adherences. Patients will need to rate their fluid and dietary adherence on a numerical rating scale which composed of 0% (None of the time) to 100% (All of the time).

SECONDARY OUTCOMES:
Feasibility of the app: interview | 12 weeks
  The feasibility of the app will be measured by the app usage. Study participants will be interviewed for app usage in term of frequency (e.g. in average how many days of usage in a week) and extent of its usage (e.g. how much time has spent on the app in a day). The intervention (mobile diet app) is consider feasible if the subject used the app more than 50% of study duration which is 42 days (6 weeks).
Acceptability: User Acceptance test (UAT) | 12 weeks
  Acceptability of the app will be measured using User Acceptance test (UAT). It consisted of 11 items and each item was rated on a 5-point Likert scale (1 = Strongly disagree, 3 = neutral, and 5 = Strongly agree).
Users Satisfaction: Likert scale | 12 weeks
  The evaluation questionnaire included 7 items evaluated using a five-point Likert scale (1 = Strongly disagree, 3 = neutral, and 5 = Strongly agree) on the composition of the app, on the design and layout of the app, and overall satisfaction.
Health Behaviour | 12 weeks
  A set of self-developed items will be used to assess the patient's perceptions of dietary adherence based on HBM constructs. Content validity have been done by 3 experts with the reported S-CVI/UA of 0.93. This part consisted of 28 items derived from available literatures, assessing different constructs of HBM
Nutrition Literacy | 12 weeks
  A dialysis-specific nutrition-related health literacy has been developed based on health literacy theory model (Sørensen et al., 2012) by the researchers and validated among HD patients with the content validity measured by S-CVI/AVE of 0.96 and construct validity measured by average variance extract (AVE) of 0.589 as well as composite reliability of 0.877 (unpublished data).
Nutritional Status | 12 weeks
  Anthropometry data will be collected by researchers at 2 time points, baseline (V0) and study end-point (V2). Malnutrition inflammation score (MIS) will be used to assess patient's nutritional status (Kalantar-Zadeh, Kopple, Block & Humphreys, 2001).
Dietary Knowledge | 12 weeks
  The kidney disease-related dietary knowledge questionnaire was modified from (Durose et al., 2004) based on the Malaysian MNT Guidelines for CKD, (MDA, 2005) which was adopted from the K-DOQI guidelines (NKF 2000; NKF 2003).

CONTACTS AND LOCATIONS:
Overall Officials: Zulfitri 'Azuan bin Mat Daud, Lecturer[Dr], Principal Investigator — Universiti Putra Malaysia; Barakatun Nisak binti Mohd Yusof, Lecturer[Dr], Principal Investigator — Universiti Putra Malaysia; Lim Jun Hao, Dietitian, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Hospital Serdang, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahmad, G., Leong, G. B., Ngo, L. Y., Meng, O. L., & Guat, L. D. (2016). 24th Report of the Malaysian Dialysis and Transplant Registry 2016. National Renal Registry Malaysia
- [Result] Campbell J, Porter J. Dietary mobile apps and their effect on nutritional indicators in chronic renal disease: A systematic review. Nephrology (Carlton). 2015 Oct;20(10):744-751. doi: 10.1111/nep.12500. PMID 25959301
- [Result] Chan YM, Zalilah MS, Hii SZ. Determinants of compliance behaviours among patients undergoing hemodialysis in Malaysia. PLoS One. 2012;7(8):e41362. doi: 10.1371/journal.pone.0041362. Epub 2012 Aug 3. PMID 22870215